CLINICAL TRIAL: NCT07108868
Title: A Phase I Dose Finding Study of MB-CART2219.1 Targeting CD19/CD22 in Adult and Pediatric Patients With Relapsed/Refractory B-cell Malignancies
Brief Title: A Phase I Dose Finding Study of MB-CART2219.1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB-CART2219.1; 2024-516838-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma; CLL; Acute Lymphoblastic Leukemia, Pediatric
Keywords: MB-CART2219.1 targeting CD19/CD22; CD19/CD22; CAR-T cells
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose finding (Experimental): Phase I dose finding and efficacy study using the 3+3 design
  Interventions: Biological: CAR-T cells targeting CD19 and CD22

INTERVENTIONS:
Biological: CAR-T cells targeting CD19 and CD22 — Using the 3+3 design, the following dose levels will be assessed:
  Dose level 1: 0.5x10e6 CAR-transduced T cells/kg; Dose level 2: 1x10e6 CAR-transduced T cells/kg; Dose level 3: 2x10e6 CAR-transduced T cells/kg; Dose level 0: 0.25x10e6 CAR-transduced T cells/kg

SUMMARY:
A Phase I dose finding study of MB-CART2219.1 targeting CD19/CD22 in adult and pediatric patients with relapsed/refractory B-cell malignancies

ELIGIBILITY:
Inclusion Criteria:

1. For Cohort I Lymphoma, adults: Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. For Cohort II ALL, pediatrics: Subject is ≥ 12 years of age at the time of signing ICF.
3. Patient or legal guardian understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
4. Able to adhere to the study visit schedule and other protocol requirements as well as agrees to continued follow up for up to 15 years as mandated by the regulatory guidelines for gene therapy trials.
5. CD19 or CD22 expression must be detected on the malignant cells by flow cytometry or immunohistochemistry. Results of previous assessments after the last treatment with CD19 targeted therapies but preceding inclusion of the patient in this trial are acceptable, if available.
6. Female Subject of childbearing potential and male subjects with female partner of childbearing potential is willing to use highly effective contraceptive methods during treatment until 12 months after IMP exposure.
7. All subjects must agree to refrain from donating blood while on study drug and for 1 year after discontinuation from this study treatment.
8. Male or female patients must have relapsed refractory (r/r) CD19 or CD22 -expressing ALL or Lymphoma/CLL and meet the following disease-specific criteria.

   1. Patients with r/r lymphoma with following entities according to 5th edition of the WHO Classification of Haematolymphoid Tumors after two or more systemic therapies, including one approved in label CAR-T-cell or bispecific antibody treatment option or with contraindications for such treatments:

      * B-lymphoblastic lymphomas
      * B-Chronic lymphocytic leukemia
      * Splenic B-cell lymphoma
      * Marginal zone lymphoma
      * Follicular lymphoma
      * Mantle cell lymphoma
      * Large B-cell lymphoma
      * Burkitt lymphoma
      * Transformation from indolent lymphoma
   2. Patients with r/r CLL after established and approved treatment options including therapy with BTK inhibitors have failed
   3. Patients with lymphoma recommended for autologous or allogeneic stem cell transplant (SCT) therapy by interdisciplinary boards, but not consenting or ineligible for this treatment (including patients with refractory disease precluding allo SCT at this time, which can be included in the study as bridge to allo SCT)
   4. Patients with lymphoma relapse after SCT, or afterCD19 or CD22 targeting therapies and with confirmed either CD19 or CD22 expression after relapse
   5. Patients with CNS involvement by lymphoma are eligible if disease is successfully controlled at the time of inclusion

Exclusion Criteria:

1. Subject received any of the following within the last 7 days of leukapheresis:

   * Any investigational agent
   * Immunsupressive medication
   * Plasmapheresis
   * Major surgery (as defined by the investigator)
   * Radiation therapy other than local therapy for underlying malignancy
   * Use of any systemic anti-neoplastic drug therapy or immune suppressive medication applied for graft versus-host-disease or other, including the use of high dose steroids e.g. >0,5 mg/kg BW methylprednisolone other than hydrocortisone replacement and other than intermittent topical, inhaled or intranasal corticosteroids which are allowed
2. Subject has ECOG > 3 at screening for inclusion in the trial
3. Subject has clinical evidence of pulmonary leukostasis, disseminated intravascular coagulation or active graft versus-host-disease
4. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or other CNS bleed, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
5. Subject has any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 500/μL
   * Absolute lymphocyte count < 200/µL at time of leukapheresis
   * Platelet count < 50,000 mm3 (platelet transfusion allowed)
   * Serum Creatinine Clearance (CrCl) < 45 mL/min
   * Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN)
   * Serum total bilirubin > 1.5 × ULN or > 3.0 mg/dL for subjects with documented Gilbert's syndrome
   * International ratio (INR) or partial thromboplastin time (PTT) > 1.5 × ULN, or history of Grade ≥ 2 hemorrhage within 30 days, or subject requires ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors)
6. Patient has no adequate vascular access for leukapheresis
7. Echocardiogram (ECHO) or multi-gated acquisition (MUGA) with left ventricular ejection fraction < 45%
8. Patient with a history of Class III or IV congestive heart failure (CHF) or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 3 months prior to starting study treatment
9. Inadequate pulmonary function defined as oxygen saturation (Sa02) < 90 % on room air
10. Subject has history of primary immunodeficiency
11. Subject is positive for human immunodeficiency virus (HIV-1), uncontrolled hepatitis B or C or active hepatitis A
12. Subject with ongoing (incl. controlled) infections or infestations where inclusion of the patient into the clinical trials may significantly jeopardize the health and wellbeing of the patient, as determined by the investigator.
13. Subject with malignancy other than the underlying malignancy in this protocol, unless this disease has been controlled for ≥ 1 year and the exception of the following noninvasive malignancies:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative
14. Patient is a female who is pregnant, nursing, or breastfeeding, or who intends to become pregnant during participation in the study
15. Patient with known hypersensitivity to any component of MB-CART2219.1 product, cyclophosphamide, fludarabine, and/or tocilizumab
16. Patient has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
17. Patient has any further condition including the presence of further laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility Phase I (CTCAE) | 6 months
  Objective: to assess feasibility, safety of ex vivo generated MB-CART2219.1 in patients with relapsed or refractory CD19 and/or CD22 positive B cell malignancies. Determination of the recommended dose of MB-CART-CD19CD22, determined on the basis of the maximum tolerated dose, defined as the highest dose level of the 2-3 dose levels tested at which <33% of patients experience DLT until d+28 after infusion of MBCART2219.1 and on the basis of the safety and efficacy data. Safety and toxicity assessment of MB-CART2219.1 per adverse events reporting classified according to CTCAE version 5.0 defined by <33% of patients experiencing DLT, or maximal administered dose. The Trial uses two separate disease and age specific cohorts for dose escalation: cohort I (Lymphoma incl. CLL, adults) and cohort II (ALL, children). For each cohort in using the standard 3+3 design, three dose levels will be assessed. Feasibility will be defined as successful treatment without major deviation from the protocol

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital , Department of Internal Medicine II, Tübingen, Baden-Wurttemberg
  - University Hospital, Clinic for Pediatric Medicine, Tübingen, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No